CLINICAL TRIAL: NCT06145438
Title: Comparing the Safety and Efficacy in the Use of Dienogest, Leuprolide Acetate, DMPA and Combined Oral Contraceptive Pills (Microgynon) on Endometriosis Patients After Conservative Surgery
Brief Title: Comparing the Safety and Efficacy in the Use of Hormonal Therapy on Endometriosis Patients After Conservative Surgery
Acronym: ENDOSafe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Yuli Trisetiyono, Principal Investigator, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000088
Record Dates: First submitted 2023-10-22; First posted 2023-11-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis Ovary
MeSH Terms: interventions — dienogest; Medroxyprogesterone Acetate; Leuprolide; Ethinyl Estradiol; Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Leuprolide Acetate (Active Comparator): Leuprolide Acetate, brand name Tapros 3.75 mg, injected intramuscularly every month for 3 months
  Interventions: Drug: Leuprolide (as Leuprolide Acetate)
- Dienogest (Experimental): Dienogest 2 mg, brand name Nelandoz 2mg, administered orally, every day for 3 months
  Interventions: Drug: Dienogest
- Depot medroxyprogesterone acetate (Experimental): Depot medroxyprogesterone acetate, brand name Depo Provera 150mg/ml, injected intramuscularly, every month for 3 months
  Interventions: Drug: Depo Medroxyprogesterone acetate
- Combined Oral Contraceptive (Experimental): Levonogestrel 150 mcg + etinilestradiol 30 mcg, brand name Mycrogynon, administered orally, every day for 3 months
  Interventions: Drug: Levonogestrel + etinilestradiol (30 mcg, brand name Mycrogynon)

INTERVENTIONS:
Drug: Dienogest — Drug is administered orally at the same time every day
  Other Names: Nelandoz
  Arms: Dienogest
Drug: Depo Medroxyprogesterone acetate — Drug is injected intramuscularly on the buttock
  Other Names: Depo Provera
  Arms: Depot medroxyprogesterone acetate
Drug: Leuprolide (as Leuprolide Acetate) — Drug is injected intramuscularly on the buttock
  Other Names: Tapros
  Arms: Leuprolide Acetate
Drug: Levonogestrel + etinilestradiol (30 mcg, brand name Mycrogynon) — Drug is administered orally at the same time every day
  Other Names: Combined oral contraceptive
  Arms: Combined Oral Contraceptive

SUMMARY:
The goal of this clinical trial is to compare safety and efficacy in endometriosis patient after conservative surgery. The main question[s] it aims to answer are:

1. Health-related quality of life (HRQoL)
2. VAS score
3. Beta estradiol
4. TNF Alpha
5. Adnexal mass recurrence

Participants will be randomized into 4 groups, each group will receive:

1. Leuprolide Acetate injection/month
2. Dienogest 2 mg/day
3. COC (mycrogynon)/day
4. DMPA injection 150mg/month Researcher will compare the efficacy and safety in the assigned group.

DETAILED DESCRIPTION:
1. Beta estradiol level is measured in the serum, before and after treatment
2. TNF alpha is measured in the serum, before and after treatment
3. Evaluation of HRQoL using the Endometriosis Health Profile-30 (EHP-30)
4. VAS score will be recorded before and after treatment
5. Adnexal massa recurrence evaluation using USG

ELIGIBILITY:
Inclusion Criteria:

Patient post surgical removal of endometriosis cyst Willing to participate

Exclusion Criteria:

1. Use of any hormonal therapy for endometriosis within the previous 16 weeks.
2. History of severe adverse drug reactions or hypersensitivity to steroid hormones.
3. Failure of previous treatment with COC, DMPA used in this study.
4. There are contraindications to the use of Leuprolide Acetate, COC, DMPA or Dienogest, such as a history or complications of thrombosis/embolism, stroke, Diabetes Mellitus, liver cirrhosis or other liver function disorders, breast, ovarian and endometrial malignancies.
5. Smoker.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
beta estradiol level | 0 and 12 weeks of treatment
  Measuring beta estradiol level on the serum
TNF alpha level | 0 and 12 weeks of treatment
  Measuring TNF alpha level on the serum

SECONDARY OUTCOMES:
VAS score | 0 and 12 weeks of treatment
  Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum. 0 means "no pain" and 10 means"worst pain
health-related quality of life (HRQoL) | 0 and 12 weeks of treatment
  Endometriosis Health Profile-30 (EHP-30). It consists of 30 items to which respondents can choose between the answers: Never (0); Rarely (1), Sometimes (2); Often (3); and Always (4). The 30 items are divided into five subscales covering 'pain', 'control and powerlessness', 'social support', 'emotional wellbeing' and 'self-image'. Each scale is standardized on a scale from 0 to 100, with lower scores indicating better QoL
Mass recurrence | 0 and 12 weeks of treatment
  Evaluate the adnexal mass using Ultrasound after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuli Trisetiyono, SpOG (K), Principal Investigator — Diponegoro University
Locations (1):
- Kariadi Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: ICF
Time Frame: Starting in March 2024
Access Criteria: Informed Consent Form will be shared to other researchers by sending email